CLINICAL TRIAL: NCT02851797
Title: Randomised, Double Blind, Placebo Controlled, Multicentre Study to Evaluate the Efficacy and Safety of Givinostat in Ambulant Patients With Duchenne Muscular Dystrophy
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of Givinostat in Ambulant Patients With Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPYDIS (DSC/14/2357/48); 2016-000401-36 (EudraCT Number)
Record Dates: First submitted 2016-07-27; First posted 2016-08-02 (Estimated); Results first posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Dystrophy; DMD; Givinostat
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — givinostat; givinostat hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- givinostat (Active Comparator): Givinostat oral suspension (10 mg/mL) twice daily
  Interventions: Drug: givinostat
- placebo (Placebo Comparator): Placebo oral suspension (10 mg/mL) twice daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: givinostat — The oral suspension of givinostat (10 mg/mL) was to be dosed in fed condition as described below:
  Givinostat or placebo starting dose
  * > or =10 and < 12.5 kg of weight: 13.3 mg bid = 1.3 ml oral suspension bid
  * > or =12.5 and < 20 kg: 16.7 mg bid =1.7 ml oral suspension bid
  * > or = 20 and < 25 kg: 20 mg bid = 2.0 ml oral suspension bid
  * > or = 25 and < 30 kg: 23.3 mg bid = 2.3 ml oral suspension bid
  * > or = 30 and < 40 kg: 26.7 mg bid = 2.7 ml oral suspension bid
  * > or = 40 and < 50 kg: 33.3 mg bid = 3.3 ml oral suspension bid
  * > or = 50 and < 60 kg: 36.7 mg bid = 3.7 ml oral suspension bid
  * > or = 60 and < 70 kg: 40 mg bid = 4 ml oral suspension bid
  * > or = 70 kg: 46.7 mg bid = 4.7 ml oral suspension bid
  Other Names: ITF2357
  Arms: givinostat
Drug: placebo — The oral suspension of placebo, manufactured to mimic givinostat, was to be dosed in fed condition as described for givinostat.
  Arms: placebo

SUMMARY:
Primary Objective

The primary objective of the study was to establish the effects of givinostat versus placebo administered chronically over 18 months to slow disease progression in ambulant DMD subjects.

Secondary Objectives

The secondary objectives of this study were:

* To assess the safety and tolerability of givinostat versus placebo administered chronically in DMD subjects
* To evaluate the PK profile of givinostat administered chronically in DMD subjects
* To evaluate the impact on quality of life (QoL) and activities of daily living of givinostat versus placebo administered chronically.

DETAILED DESCRIPTION:
This was a phase 3, randomised, double-blind, placebo-controlled, multicentre study to evaluate the efficacy and safety of givinostat in ambulant subjects with DMD. This study included ambulant male paediatric subjects aged ≥ 6 years at baseline affected by DMD.

A total of 179 male ambulant subjects was randomized 2:1 (givinostat: placebo).

Subjects were stratified for their concomitant use of steroids in 4 strata:

1. Deflazacort daily regimen
2. Deflazacort intermittent regimen
3. Other steroids daily regimen
4. Other steroids intermittent regimen. The study duration was planned to be 19 months.

Givinostat or placebo oral suspension (10 mg/mL) was administered orally as 2 oral doses daily while the subject were in fed state, according to the child's weight.

Study drug should have been permanently stopped if any of the following occurred:

* severe drug-related diarrhoea;
* any drug-related Serious Adverse Event;
* QTcF >500 msec;
* platelets count ≤50 x 10^9/L.
* white blood cells ≤2.0 x 10^9/L
* hemoglobin ≤8.0 g/dL

Study drug should have been temporarily stopped if any of the following occurred:

* moderate or severe diarrhoea.
* platelets count <75 x 10^9/L but >50 x 10^9/L (the treatment should been temporarily stopped and a platelets count was to be performed and re-tested until platelets normalized);
* white blood cell <3.0 x 10^9/L but >2.0 x 10^9/L (the treatment should be temporarily stopped and white blood cells had to be measured by 1 week and re-tested until white blood cells normalized);
* hemoglobin <10.0 g/dL but > 8.0 g/dL (the treatment should be temporarily stopped and hemoglobin had to be measured by 1 week and re-tested until hemoglobin normalized);
* Triglycerides >300 mg/dL (3.42 mmol/L) in fasting condition (the treatment should be temporarily stopped and triglycerides measured every 2 weeks until triglycerides returned to levels below 300mg/dL (3.42 mmol/L)

In case the study drug was temporarily stopped, the study drug could be resumed at a level 20% smaller than the one at which the Adverse Event leading to temporary stop occurred, once platelets and/or white blood cell and/or hemoglobin normalized and/or triglycerides returned to levels below 300 mg/dL (3.42 mmol/L) or diarrhoea was mild.

In addition, in case a subject had a consistent (e.g., at least 2 consecutive evaluations) platelets count ≤150 x 10^9/L and didn't meet the stopping criteria for platelets, the Investigator should have to reduce the dose by 20% of the current dose.

Only one dose reduction was allowed during the treatment period.

This trial design a single planned interim analysis. The interim was governed by an IDMC in order to solely assess futility.

ELIGIBILITY:
Inclusion Criteria:

1. Are an ambulant male aged ≥6 years at randomisation with DMD characteristic clinical symptoms or signs (e.g., proximal muscle weakness, Gowers' maneuver, elevated serum creatinine kinase level) already present at screening;
2. Have DMD diagnosis confirmed by genetic testing;
3. Are able to give informed assent and/or consent in writing signed by the subject and/or parent/legal guardian (according to local regulations);
4. Are able to complete 2 Four Stairs Climb test (4SC) screening assessments; the results of these tests must be within ±1 second of each other;
5. Have the mean of 2 screening 4SC assessments ≤8 seconds;
6. Have time to rise from floor between ≥3 and <10 seconds at screening
7. Have manual muscle testing (MMT) of quadriceps at screening Grade ≥- 3;
8. Have used systemic corticosteroids for a minimum of 6 months immediately prior to the start of study treatment, with no significant change in corticosteroids type or dosage or dosing regimen (excluding changes related to body weight change) for a minimum of 6 months immediately prior to start of study treatment and a reasonable expectation that dosage and dosing regimen will not change significantly for the duration of the study.
9. Subjects must be willing to use adequate contraception.

Exclusion Criteria:

1. Have exposure to another investigational drug within 3 months prior to the start of study treatment;
2. Have exposure to idebenone within 3 months prior to the start of study treatment;
3. Have exposure to any dystrophin restoration product (e.g., Ataluren, Exon skipping) within 6 months prior to the start of study treatment;
4. Use of any pharmacologic treatment, other than corticosteroids, that might have had an effect on muscle strength or function within 3 months prior to the start of study treatment (e.g., growth hormone); Vitamin D, calcium, and any other supplements will be allowed as long as their intake has been stable for 3 months prior to the start of study treatment; Testosterone will also be allowed if it is used as a replacement therapy for the treatment of delayed puberty, and testosterone dose and regimen have been stable for at least 6 months and circulating testosterone levels are within the normal ranges for the subject's age;
5. Have surgery that might have an effect on muscle strength or function within 3 months before study entry or planned surgery at any time during the study;
6. Loss of ≥30 degrees of plantar flexion from the normal range of movement at the ankle joint due to contracture (i.e. fixed loss of more than 10 degrees of plantar flexion from plantigrade, assuming normal range of dorsiflexion of 20 degrees;
7. Change in contracture treatment such as serial casting, contracture control devices, night splints, stretching exercises (passive, active, self) within 3 months prior to enrollment, or expected need for such intervention during the study;
8. Have presence of other clinically significant disease, which, in the Investigator's opinion, could adversely affect the safety of the subject, making it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results;
9. Have a diagnosis of other uncontrolled neurological diseases or presence of relevant uncontrolled somatic disorders that are not related to DMD;
10. Have platelets count at screening < Lower Limit of Normal (LLN);
11. Have symptomatic cardiomyopathy or heart failure (New York Heart Association Class III or IV) or left ventricular ejection fraction <50% at screening;
12. Have a current or history of liver disease or impairment;
13. Have inadequate renal function, as defined by serum Cystatin C >2 x the upper limit of normal (ULN);
14. Have Triglycerides > 300 mg/dL (3.42 mmol/L) in fasting condition at screening visit;
15. Have a positive test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus at screening15.
16. Have a baseline QTcF >450 msec, or history of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, or family history of long QT syndrome);
17. Have a psychiatric illness/social situations rendering the potential subject unable to understand and comply with the muscle function tests and/or with the study protocol procedures;
18. Have any hypersensitivity to the components of study medication;
19. Have a sorbitol intolerance or sorbitol malabsorption, or have the hereditary form of fructose intolerance.
20. Have contraindications to MRI or MRS (e.g., claustrophobia, metal implants, or seizure disorder).

At the discretion of the Investigator, subjects not meeting inclusion/exclusion criteria may be re-screened twice with an interval of at least 3 months between assessments.

Ages: 6 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — to take part in the study, subjects should be:
  1) ambulant males aged ≥ 6 years at randomization with DMD-characteristic clinical symptoms or signs (eg, proximal muscle weakness, Gowers' maneuver, elevated serum creatinine kinase level) already present at screening, 2. should have a DMD diagnosis confirmed by genetic testing
Enrollment: 179 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Mercuri, MD, PhD, Principal Investigator — Istituto di Ricovero e Cura a Carattere Scientifico, IRCCS
Locations (42):
- United States (13):
  - Neuromuscular Research Center UC Davis Department of Physical Medicine and Rehabilitation, Davis, California
  - Rady Children's Hospital center - UCSD Department of Neuroscience, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center - Division Neurology, Hartford, Connecticut
  - Child Health Research Institute - Department of Pediatrics, Gainesville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - MD Rare Disease Research, LLC, Atlanta, Georgia
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - University of Minnesota - Department of Neurology, Minneapolis, Minnesota
  - Washington University School of Medicine in St Louis - Department of Neurology, St Louis, Missouri
  - Shriners Hospitals for Children, Portland, Oregon
  - The Children's Hospital of Philadelphia Colket Translational Research Building, Philadelphia, Pennsylvania
  - Virginia Commonwealth University Childrens Hospital of Richmond at Virginia Commonwealth University, Richmond, Virginia
- Belgium (2):
  - University Hospitals Leuven, Neuromuscular Reference Centre, Child Neurology, Leuven
  - Hospital de La Citadelle, Centre de Référence des Maladies Neuromuscolaires (CRMN), Liège
- Canada (3):
  - Kinsmen Research Centre - Alberta Children's Hospital - Alberta Health Services, Calgary, Alberta
  - The University of British Columbia, Children's and Womens Health Centre of BC Branch, Vancouver, British Columbia
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario
- France (2):
  - CHU de Nantes - Hotel-Dieu - Hopital Nord Laennec, rez-de-chausse haut ail Ouest, Nantes
  - Hopital Armand Trousseau I-Motion, Plateforme d'essais cliniques pédiatriques, Paris
- Germany (3):
  - Universitatsklinikum Essen - Kinder und Jugendmedizin Neuropadiatrie, Essen
  - Klinik un Policlinik fur Kinder und Jugendmedizin - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Klinikum der Uniersitat Munchen - Campus Innenstadt, München
- Institute of Neurology - Schneider Children's Medical Center of Israel Kaplan, 14, Petah Tikva, Israel
- Italy (7):
  - IRCCS Istituto G.Gaslini, U.O.S.D. Centro Traslazionale di Miologia e Patologie Neurodegenerative, Genova
  - A.O.U. Policlinico G. Martino, U.O.C. Neurologia e Malattie Neuromuscolari, Messina
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, UOS di Neurologia Pediatrica, Milan
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Centro Clinico NeMO Fondazione Serena ONLUS Area SUD, Milan
  - Ospedale Pediatrico Bambin Gesù, Malattie Neuromuscolari e Neurodegenerative, Roma
  - Fondazione Policlinico Universitario "A.Gemelli", UOC Neuropsichiatria Infantile, Roma
- Netherlands (2):
  - Leiden University Medical Center LUMC, Leiden
  - Radboud University Medical Centre, Nijmegen
- Clinic of Neurology and Psychiatry for Children and Youth - Neurology Department Dr. Subotic 6a,, Belgrade, Serbia
- Spain (4):
  - Hospital Sant Joan de Déu - Neuromuscular Pathology Unit, Esplugues de Llobregat, Barcelona
  - Hospital Materno-Infantil - Passeig de la Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politécnic de la Fe - Servicio Neurologia, Valencia
- United Kingdom (4):
  - Alder Hey Children's Hospital NHS Trust, Liverpool
  - UCL Great Ormond Street Institute of Child Health, Dubowitz Neuromuscular Centre and MRC Centre for NMD, London
  - The John Walton Muscular Dystrophy Research Centre - Freeman Hospital - Newcastle University - Institute of Genetic Medicine, Newcastle upon Tyne
  - The Robert Jones and Agnes Hunt Orthopaedic Hospital - NHS Foundation Trust, Oswestry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mercuri E, Vilchez JJ, Boespflug-Tanguy O, Zaidman CM, Mah JK, Goemans N, Muller-Felber W, Niks EH, Schara-Schmidt U, Bertini E, Comi GP, Mathews KD, Servais L, Vandenborne K, Johannsen J, Messina S, Spinty S, McAdam L, Selby K, Byrne B, Laverty CG, Carroll K, Zardi G, Cazzaniga S, Coceani N, Bettica P, McDonald CM; EPIDYS Study Group. Safety and efficacy of givinostat in boys with Duchenne muscular dystrophy (EPIDYS): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Neurol. 2024 Apr;23(4):393-403. doi: 10.1016/S1474-4422(24)00036-X. PMID 38508835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Within the overall population, a total of 118 subjects were enrolled in the givinostat group. A total of 61 subjects were enrolled in the placebo group.
Groups:
- Givinostat: Givinostat oral suspension (10 mg/mL) twice daily
  givinostat: The oral suspension of givinostat (10 mg/mL) was to be dosed in fed condition as described below: Givinostat or placebo starting dose
  * > or =10 and < 12.5 kg of weight: 13.3 mg bid = 1.3 ml oral suspension bid
  * > or =12.5 and < 20 kg: 16.7 mg bid =1.7 ml oral suspension bid
  * > or = 20 and < 25 kg: 20 mg bid = 2.0 ml oral suspension bid
  * > or = 25 and < 30 kg: 23.3 mg bid = 2.3 ml oral suspension bid
  * > or = 30 and < 40 kg: 26.7 mg bid = 2.7 ml oral suspension bid
  * > or = 40 and < 50 kg: 33.3 mg bid = 3.3 ml oral suspension bid
  * > or = 50 and < 60 kg: 36.7 mg bid = 3.7 ml oral suspension bid
  * > or = 60 and < 70 kg: 40 mg bid = 4 ml oral suspension bid
  * > or = 70 kg: 46.7 mg bid = 4.7 ml oral suspension bid
Period: Overall Study
Arm/Group | Givinostat | Placebo
Started | 118 | 61
All Enrolled Subjects | 118 | 61
ITT Population | 118 | 61
Safety Set | 118 | 61
PK Analysis Set | 117 | 0
Target Population | 81 | 39
MR Cohort | 77 | 37
Completed | 111 | 59
Not Completed | 7 | 2
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Population: Number of Subjects Enrolled in Each Country (Overall Population).The all-enrolled subjects set included all subjects who were randomised to study treatment. The overall all-enrolled subjects set included all subjects in both the target and off-target populations (Group A + Group B) who were randomised to study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Givinostat | Placebo | Total
Number analyzed (Participants) | 118 | 61 | 179
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 118 | 61 | 179
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.78 (2.022) | 9.97 (2.082) | 9.84 (2.039)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 118 | 61 | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 3 | 12
  Not Hispanic or Latino | 109 | 58 | 167
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 106 | 57 | 163
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 6 | 15
  Netherlands | 5 | 3 | 8
  Belgium | 6 | 3 | 9
  United States | 24 | 19 | 43
  Italy | 24 | 13 | 37
  United Kingdom | 10 | 3 | 13
  Israel | 1 | 0 | 1
  France | 9 | 5 | 14
  Serbia | 0 | 1 | 1
  Germany | 13 | 2 | 15
  Spain | 17 | 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in 4 Standard Stairs (4SC) Climb After 18 Months of Treatment
Description: The time (in seconds) to climb 4 standard-sized stairs is a TFT that represents stair-climbing ability. The test was evaluated by qualified functional evaluators (ie, physiotherapists) who were different from the site personnel who reviewed subjects' safety results. The test was performed in a standardised manner described in a specific site manual. Baseline 4SC was the measurement taken at the randomization assessment, unless this was missing, in which case baseline was taken as the last non missing value recorded prior to or on the date of first study treatment. The shorter the time, the better the outcome.
Time Frame: Baseline and 18 months
Population: ITT analysis set: the intent-to-treat (ITT) analysis set included all subjects who were randomised, received at least one dose of study drug, and had at least 1 non-missing post-baseline 4SC measure or missing post-baseline 4SC measure due to being either non-ambulatory or otherwise physically unable to perform the assessment, irrespective of any deviation from the protocol or premature discontinuation.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 81 | 39
seconds | 1.27 (0.040) | 1.48 (0.058)
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Log transformation applied; Test type: Superiority — LS Means, CIs, and p-values are obtained from an analysis of covariance (ANCOVA) model on change from baseline in 4SC at Month 18 with baseline values for: 4SC, time to rise from floor, time to run/walk 10 metres, distance walked in 6 minutes and re-derived age at first dose fitted as covariates, with concomitant steroid use and treatment group as independent classification factors; p = 0.0345, ANCOVA — LS Means, CIs, and p-values are obtained from ANCOVA model on change from baseline in 4SC at Month 18 with baseline values for: the above mentioned parameters as covariates, with steroid use and treatment group as independent classificat factors; generalised least square mean ratio = 0.86, 95% CI 2-sided [0.745 to 0.989] — LS Means, CIs, and p-values are obtained from ANCOVA model on change from baseline in 4SC at Month 18 with baseline values for: the above mentioned parameters as covariates, with steroid use and treatment group as independent classificat factors

2. Secondary Outcome: Mean Change From Baseline in Time to Rise From Floor After 18 Months of Treatment
Description: An analysis of time (in seconds) to rise from the floor by change from baseline at 18 months is presented for the Target Population in the ITT analysis set. The shorter the time, the better the outcome.
Time Frame: Baseline and 18 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 81 | 39
seconds | 9.33 [5.821 to 12.838] | 12.61 [7.491 to 17.724]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Test type: Superiority — LS Means, CIs, and p-values are obtained from an analysis of covariance (ANCOVA) model on change from baseline in time to rise from the Floor at Month 18 with baseline values for: 4SC, time to rise from floor, time to run/walk 10 m, distance walked in 6 minutes and re-derived age at first dose fitted as covariates, with concomitant steroid use and treatment group as independent classification factors; p = 0.3044, ANCOVA — See comment above; difference in least square means = -3.28, 95% CI 2-sided [-9.573 to 3.018] — See comment above

3. Secondary Outcome: Mean Change From Baseline in the Six-minute Walking Test (6MWT) After 18 Months of Treatment
Description: This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes.
  The 6-Minute Walk Test is a useful measure of functional capacity targeted at people with at least moderately severe impairment. A modified version of the 6MWT recommended by American Thoracic Society (2002) for use in adults was performed.
  The longer the walked distance the better the outcome.
Time Frame: Baseline and 18 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: meters
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 81 | 39
meters | -38.43 [-50.704 to -26.153] | -48.38 [-66.288 to -30.482]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Test type: Superiority — LS Means, CIs, and p-values are obtained from an analysis of covariance (ANCOVA) model on change from baseline in distance walked at the end of the 6-minute walking test (6MWT) at Month 18 with baseline values for: 4SC, time to rise from floor, time to run/walk 10 metres, distance walked in 6 minutes and re-derived age at first dose fitted as covariates, with concomitant steroid use and treatment group as independent classification factors; p = 0.3723, ANCOVA — See comment above; LS means, CIs, p-values were obtained from analysis of covariance model on change from baseline in distance walked at the end of the 6MWT at Month18; Difference in least square means = 9.96, 95% CI 2-sided [-12.071 to 31.983] — See comment above

4. Secondary Outcome: Mean Change From Baseline in Total North Star Ambulatory Assessment (NSAA) Score After 18 Months of Treatment
Description: The total North Star Ambulatory Assessment (NSAA) is a 17-item rating scale that is used to measure functional motor abilities in ambulant children with Duchenne Muscular Dystrophy (DMD). It is usually used to monitor the progression of the disease and treatment effects. The 17 items of the NSAA, ranging from standing to running 10 meters, were graded using the standard score card with each assessment rated as 0 - unable to achieve independently, 1 - modified method but achieves goal independent of physical assistance from another, or 2 - normal with no obvious modification of activity. This scale is ordinal with 0 as the minimum score (indicating full disfunctionality, i.e. the worst outcome) and with 34 as the maximum score indicating fully-independent function (the best outcome).
Time Frame: Baseline and 18 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 81 | 39
score on a scale | -2.66 [-3.563 to -1.759] | -4.58 [-5.891 to -3.260]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Test type: Superiority — LS Means, CIs, and p-values are obtained from an analysis of covariance (ANCOVA) model on change from baseline in total NSAA score at Month 18 with baseline values for: total NSAA score, 4SC, time to rise from floor, time to run/walk 10 metres, distance walked in 6 minutes and re-derived age at first dose fitted as covariates, with concomitant steroid use and treatment group as independent classification factors; p = 0.0209, ANCOVA — Same comment as above; Difference in least square means = 1.91, 95% CI 2-sided [0.295 to 3.533] — Same comment as above

5. Secondary Outcome: Cumulative Loss of Function on the NSAA
Description: Subject cumulative number of failures across all postbaseline visits was the endpoint of interest for analysis.
  For each subject at each postbaseline visit, failure to perform each of the 17 items of the NSAA was assessed, where "failure" was defined as a score transition from 2 or 1 at baseline to 0 at the respective visit. The total number of failed items for the visit was calculated (maximum of 17 failed items per visit per subject). The subject's cumulative number of failures across all visits was the sum of the total failures at each postbaseline visit.
Time Frame: over 18 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: cumulative number of failures
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 81 | 39
cumulative number of failures | 3.42 [2.692 to 4.334] | 5.56 [4.002 to 7.715]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Test type: Superiority — Estimated cumulative failures, ratio of cumulative failures, CIs, and p-values are obtained from a negative binomial regression on the subject cumulative number of failures across all post-baseline visits. Total failed items at baseline, baseline values for: 4SC, time to rise from floor, time to run/walk 10 metres, distance walked in 6 minutes and re-derived age at first dose were included as independent covariates, with treatment group and steroid use included as indep classification factors; p = 0.0202, negative binomial regression model — same comment as above; Estimated cumulative failures, their ratio were obtained from a negative binomial regression on the cumulative N of failures across all visits; Ratio of cumulative failures = 0.61, 95% CI 2-sided [0.408 to 0.927] — A lower ratio indicates a greater reduction in cumulative loss of function across 18 months for givinostat compared with placebo. See also comment above

6. Secondary Outcome: Mean Change From Baseline of Muscle Strength Normalized Overtime
Description: The mean change of muscle strength normalized was evaluated by knee extension and elbow flexion normalized by subject weight, both measured by hand-held myometry (HHM).
Time Frame: Baseline and 18 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Newtons/kg
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 81 | 39
Newtons/kg
  Overall knee extension | -0.32 [-0.441 to -0.197] | -0.50 [-0.681 to -0.328]
  Overall elbow flexion | -0.10 [-0.174 to -0.031] | -0.19 [-0.292 to -0.085]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Overall knee extension; Test type: Superiority — LS Means, CIs, and p-values are obtained from an analysis of covariance (ANCOVA) model on change from baseline in normalised muscle strength at Month 18 with baseline normalised muscle strength and re-derived age at first dose fitted as covariates, with concomitant steroid use and treatment group as independent classification factors; p = 0.0902, ANCOVA — same comment as above; Difference in least square means = 0.19, 95% CI 2-sided [-0.030 to 0.401] — same comment as above
Statistical Analysis 2: Comparison: Givinostat vs Placebo; Overall elbow flexion; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.1818, ANCOVA — same comment as above; Difference in least square means = 0.09, 95% CI 2-sided [-0.041 to 0.213] — same comment as above

7. Secondary Outcome: Mean Change From Baseline in Vastus Lateralis Muscle Fat Fraction (VL MFF) at 18 Months
Description: Vastus lateralis muscle fat fraction (VL MFF) was expressed as fat infiltration in this muscle. Fat infiltration was assessed by Magnetic Resonance (MRS).
Time Frame: Baseline and 18 months
Population: MR cohort: the MR cohort included all subjects in the Target Population who were randomised to study treatment and completed at least one post-baseline MRI/MRS assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of fat
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 77 | 37
percentage of fat | 7.63 [6.098 to 9.172] | 10.56 [8.331 to 12.783]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Test type: Superiority — LS Means, CIs, and p-values are obtained from an analysis of covariance (ANCOVA) model on change from baseline in VL MFF at Month 18 with baseline VL MFF and re-derived age at first dose fitted as covariates, with concomitant steroid use and treatment group as independent classification factors; p = 0.0354, ANCOVA — Same comment as above; Difference in least square means = -2.92, 95% CI 2-sided [-5.641 to -0.204] — Same comment as above

8. Secondary Outcome: Number of Subjects Experiencing Treatment-emergent AEs (TEAEs), Serious AEs (SAEs), Mild TEAE Moderate TEAE, Severe TEAE
Description: Adverse Events are unfavorable changes in health, including abnormal laboratory findings, that occur in trial participants during the clinical trial or within a specified period following the trial.
  Serious Adverse Events include adverse events that result in death, require either inpatient hospitalization or the prolongation of hospitalization, are life-threatening, result in a persistent or significant disability/incapacity or result in a congenital anomaly/birth defect. Other important medical events, based upon appropriate medical judgment, may also be considered Serious Adverse Events if a trial participant's health is at risk and intervention is required to prevent an outcome mentioned.
Time Frame: Baseline through end of study, that is the end of 18° month
Population: SAF analysis set: the safety analysis set included all subjects who were randomized and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 118 | 61
Participants
  Subjects with TEAE | 112 | 57
  Subjects with serious AE | 8 | 2
  Subjects with mild AE | 69 | 39
  Subjects with moderate AE | 38 | 17
  Subjects with severe AE | 5 | 1

9. Secondary Outcome: Evaluation of Acceptability/Palatability of the Oral Suspension
Description: Acceptability and palatability of the oral suspension over time are presented. More in details, child perception of the medicine at the three timepoints hereunder specified; parent perception of the medicine based on the child's reaction at the same three timepoints; and parent problems administering the medication at the same timepoints are reported.
Time Frame: Week 4, EOS, early withdrawal
Population: SAF analysis set: the safety analysis set included all subjects who were randomised and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 118 | 61
Participants
  Child perception - week 4 - dislike very much | 31 | 11
  Child perception - week 4 - dislike a little | 21 | 17
  Child perception - week 4 - not sure | 30 | 16
  Child perception - week 4 - like a little | 19 | 12
  Child perception - week 4 - like very much | 11 | 3
  Child perception - EOS - dislike very much | 21 | 7
  Child perception - EOS - dislike a little | 24 | 13
  Child perception - EOS - not sure | 34 | 16
  Child perception - EOS - like a little | 19 | 10
  Child perception - EOS - like very much | 7 | 9
  Child perception - early withdrawal - dislike very much | 1 | 0
  Child perception - early withdrawal - dislike a little | 1 | 0
  Child perception - early withdrawal - not sure | 2 | 0
  Child perception - early withdrawal - like a little | 1 | 0
  Child perception - early withdrawal - like very much | 0 | 0
  Parent perception - week 4 - unpleasant | 50 | 31
  Parent perception - week 4 - not sure | 28 | 10
  Parent perception - week 4 - pleasant | 35 | 18
  Parent perception - EOS - unpleasant | 42 | 14
  Parent perception - EOS - not sure | 40 | 22
  Parent perception - EOS - pleasant | 26 | 19
  Parent perception - early withdrawal - unpleasant | 1 | 0
  Parent perception - early withdrawal - not sure | 3 | 0
  Parent perception - early withdrawal - pleasant | 1 | 0
  Parent admin problems - week 4 - yes | 6 | 1
  Parent admin problems - week 4 - no | 107 | 58
  Parent admin problems - EOS - yes | 5 | 0
  Parent admin problems - EOS - no | 102 | 55
  Parent admin - early withdrawal - yes | 0 | 0
  Parent admin - early withdrawal - no | 5 | 0

ADVERSE EVENTS:
Time Frame: Throughout the study till the end of study (month 18, visit 15). More precisely at Visits 4 and 7 (month 1), at Visit 9 (month 2), at Visit 10 (month 3), at Visit 11 (month 6), at Visit 12 (month 9), at Visit 13 (month 12), at Visit 14 (month 15), at Visit 15 (EOS, month 18) and at the FUV (Follow-Up Visit to be performed after 4 weeks from the last dose of study drug (ie, 4 weeks ± 7 days)).
Arm/Group | Givinostat | Placebo
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/61
Serious Adverse Events (participants affected / at risk) | 8/118 | 2/61
Other Adverse Events (participants affected / at risk) | 112/118 | 57/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Givinostat (N=118) | Placebo (N=61)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Givinostat (N=118) | Placebo (N=61)
Diarrhoea (Gastrointestinal disorders) | 43 (117) | 11 (16)
Vomiting (Gastrointestinal disorders) | 34 (64) | 8 (12)
Abdominal pain (Gastrointestinal disorders) | 25 (52) | 9 (16)
Abdominal pain upper (Gastrointestinal disorders) | 17 (21) | 7 (9)
Nausea (Gastrointestinal disorders) | 8 (9) | 4 (6)
Constipation (Gastrointestinal disorders) | 8 (9) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 31 (50) | 19 (27)
Upper respiratory tract infection (Infections and infestations) | 7 (9) | 8 (9)
Rhinitis (Infections and infestations) | 6 (11) | 7 (8)
Gastroenteritis (Infections and infestations) | 9 (12) | 3 (3)
Ear infection (Infections and infestations) | 3 (5) | 4 (4)
Influenza (Infections and infestations) | 3 (3) | 4 (4)
Platelet count decreased (Investigations) | 51 (82) | 9 (14)
Blood triglycerides increased (Investigations) | 14 (19) | 3 (6)
Fall (Injury, poisoning and procedural complications) | 15 (24) | 13 (18)
Contusion (Injury, poisoning and procedural complications) | 11 (32) | 3 (6)
Ligament sprain (Injury, poisoning and procedural complications) | 8 (9) | 3 (4)
Limb Injury (Injury, poisoning and procedural complications) | 6 (8) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (14) | 7 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (9) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (18) | 2 (2)
Headache (Nervous system disorders) | 28 (41) | 14 (30)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 9 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (21) | 5 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 1 (1)
Pyrexia (General disorders) | 15 (18) | 5 (6)
Fatigue (General disorders) | 9 (10) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 11 (18) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 14 (22) | 1 (3)
Decreased appetite (Metabolism and nutrition disorders) | 8 (10) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 19 (27) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 11 (14) | 4 (4)
Cardiac disorders (Cardiac disorders) | 8 (12) | 1 (2)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 6 (11) | 3 (4)
Eye disorders (Eye disorders) | 5 (8) | 4 (4)
Vascular disorders (Vascular disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT02851797/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT02851797/SAP_001.pdf